CLINICAL TRIAL: NCT01815372
Title: Ultrasound-guided Nerve Blocks for the Sciatic and Saphenous Nerves: Characteristics of the Single Penetration Dual Injection (SPEDI) Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Jens Borglum Neimann, Consultant anesthetist, PhD, Ass. Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPEDI
Record Dates: First submitted 2012-11-26; First posted 2013-03-21 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Lower Leg Surgery, e.g. Ankle Fractures
Keywords: nerve blocks; ultrasound-guided; leg surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPEDI (Experimental): These are the patients that will be randomized to receive a SPEDI block of the sciatic and saphenous nerve with at single needle penetration of the skin
  Interventions: Procedure: Single penetration dual injection (SPEDI) block technique to block the sciatic and the saphenous nerve with one needle penetration of the skin
- Popliteal sciatic and mid-femoral saphenous (Active Comparator): These are the patients that will be randomized to the administration of a popliteal sciatic nerve block combined with a mid-femoral saphenous nerve block with two separate injections
  Interventions: Procedure: The classical popliteal sciatic nerve block combined with the mid-femoral saphenous nerve block

INTERVENTIONS:
Procedure: Single penetration dual injection (SPEDI) block technique to block the sciatic and the saphenous nerve with one needle penetration of the skin
  Arms: SPEDI
Procedure: The classical popliteal sciatic nerve block combined with the mid-femoral saphenous nerve block
  Arms: Popliteal sciatic and mid-femoral saphenous

SUMMARY:
Background and aims: Ultrasound-guided (USG) nerve blocks of the sciatic nerve (popliteal level = PL) and the saphenous nerve (mid-femoral level = MFL) provides analgesia following leg surgery. Traditionally two separate injections are performed. The aim was to describe a novel, faster USG block combination requiring only one skin penetration to block the sciatic and saphenous nerves; i.e. the SPEDI block = Single PEnetration Dual Injection.

Methods: A randomized, controlled and double-blinded trial. Following ethics committee approval 60 patients will be randomized to the administration of an USG SPEDI block compared to two separate USG blocks of the saphenous (MFL) and sciatic (PL) nerves. Blocks will be performed after induction of general anaesthesia. Outcome measures will be performance time (primary outcome measure), Post-Anaesthesia Care Unit pain scores (VAS scores 0-10), block difficulty level (easy, middle, difficult), opioid consumption (in the PACU), serum-ropivacaine pharmacokinetics (blood sample 0-180 minutes). Both block combinations will be evaluated by MR imaging (MRI).

Hypothesis: The USG SPEDI block combination is expected to be performed significantly faster without moving the leg, and achieve successful perioperative pain management. The SPEDI block may find important use in the emergency setting.

ELIGIBILITY:
Inclusion Criteria:

* lower leg surgery
* American Society of Anesthesiologist (ASA) score I-III
* Can cooperate in the study
* Speaks and understand the Danish language
* General anesthesia

Exclusion Criteria:

* Intake of oral morphine above 40 mg per day
* Know allergy to ropivacaine
* Abuse of alcohol or other substance abuse
* Neuropathy
* Pregnant
* Nerve block contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Performance time (seconds and minutes). Time measurement from the time the ultrasound transducer is placed on the skin and until the needle is taken out of the body. | The measurement (seconds and minutes) will take place in the operating room. This will normally be within a time frame of 1 minute to 10 minutes.
  The time measurement is done with a normal clock - measuring seconds and minutes.

SECONDARY OUTCOMES:
Pain score (VAS score 0-10). | When the patient are evaluated in the recovery unit upon arrival and when the patient is discharged from the recovery unit. This means from time 0 hours (arrival in the PACU) and normally until 2 hours after arrival in the PACU.
Sensory dermatome testing. | Normally until 2 hours postoperatively.
  Sensory dermatome testing is done with cold ethanol on skin test. All dermatomes on the leg and foot are tested, and there is a comparison of the outcome between the operated leg and the not-operated leg.

OTHER OUTCOMES:
Opioid consumption (micrograms of sufentanil) in total in the recovery unit. | Normally from 0 hours until 2 hours after arrival in the recovery unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark